CLINICAL TRIAL: NCT01904006
Title: Improvement of Live Birth Rate With a New Standardized Human Embryo Culture System: a Prospective, Randomized, Controlled Trial
Brief Title: Impact of Human Embryo Culture System on Live Birth
Acronym: AGRUPADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVISEV-003AGR
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Embryo Culture
Keywords: grouped embryo culture; embryo density; low oxygen; benchtop incubator; culture condition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Culture Condition (Experimental): Intervention group embryos cultured grouped under low oxygen tension in benchtop incubators.
  Interventions: Procedure: New Culture Condition
- Standard Culture Condition (Active Comparator): Control group embryos cultured individually under atmospheric oxygen tension in large-box incubators.
  Interventions: Procedure: Standard Culture Condition

INTERVENTIONS:
Procedure: New Culture Condition — Intervention group embryos cultured grouped (5 embryos per drop) under low oxygen tension (5%) in benchtop incubators.
  Arms: New Culture Condition
Procedure: Standard Culture Condition — Control group embryos cultured individually (1 embryo per drop) under atmospheric oxygen tension (20%) in large-box incubators.
  Arms: Standard Culture Condition

SUMMARY:
Previous studies in human and different mammals have proved that the embryo group culture (in the same culture medium drop) using a reduced volume is associated with a better embryo development. This is due to the effect of different autocrine and paracrine factors secreted by the embryos. Besides, previous studies with embryos from human and other mammals have shown that a high oxygen concentration may have a negative effect on embryo quality due to the generation of reactive oxygen species, which cause oxidative stress. The embryo culture at low oxygen tension is correlated to better success rates in IVF/ICSI treatments.

The purpose of this study is to evaluate the combined effect of the embryo group culture and the low oxygen tension on the embryo development and the results of the IVF/ICSI treatments. The specific goal is to compare the embryo group culture in a reduced volume of medium at a low oxygen tension (5%) with the standard individual culture at an atmospheric oxygen tension (20%). The first culture condition will be applied in a K-MINC incubator (COOK Medical®), whereas the second condition will be applied using a Heracell incubator (Heraeus®).

ELIGIBILITY:
Inclusion Criteria:

* <38 years (with own oocytes) / <45 years (with oocyte donation).
* First treatment with own oocytes / any treatment with oocyte donation.
* ≥10 oocytes with a diameter of ≥10 mm.

Exclusion Criteria:

* Diseases that affect endometrial receptivity: endometriosis, hydrosalpinx, ovarian hyperstimulation syndrome, obesity, endocrinopathies, thrombophilia, congenital or acquired uterine anomalies.
* Patients under a treatment with genetic preimplantation diagnosis.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | April 2013 - October 2016
  Confirmed when a gestational sac with heartbeat was observed in the uterus by ultrasound examination, performed 2-3 weeks after the positive result of the beta-hCG pregnancy test.

SECONDARY OUTCOMES:
Implantation rate | April 2013 - October 2016
  Number of embryos implanted per number of embryos transferred
Live birth rate | April 2013 - October 2016
  Number of newborns per pregnancy achieved

OTHER OUTCOMES:
Fecundation rate | April 2013 - October 2016
Mean number of viable embryos | April 2013 - October 2016
Blastocyst rate | April 2013 - October 2016
Mean number of embryos transferred | April 2013 - October 2016
Live Birth rate per embryos transferred | April 2013 - October 2016
Multiple pregnancy rate | April 2013 - October 2016
Clinical miscarriage rate | April 2013 - October 2016

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Ruiz, MSc, Study Chair — Vida Recoletas Sevilla; Victor Blasco, MSc, Study Chair — Vida Recoletas Sevilla; Manuel Fernandez-Sánchez, PhD, Study Director — Vida Recoletas Sevilla
Locations (1):
- IVI Sevilla, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruiz M, Santamaria-Lopez E, Blasco V, Hernaez MJ, Caligara C, Pellicer A, Fernandez-Sanchez M, Prados N. Effect of Group Embryo Culture under Low-Oxygen Tension in Benchtop Incubators on Human Embryo Culture: Prospective, Randomized, Controlled Trial. Reprod Sci. 2020 Jul;27(7):1522-1533. doi: 10.1007/s43032-020-00150-5. Epub 2020 Jan 28. PMID 31994003